CLINICAL TRIAL: NCT02717910
Title: Digital Health Game as an Intervention Supporting Tobacco-related Health Literacy in Early Adolescents: a Feasibility Study
Brief Title: Digital Health Game as an Intervention Supporting Tobacco-related Health Literacy in Early Adolescents
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Turku (Other)
Responsible Party: Principal Investigator, Heidi Parisod, Doctoral candidate, MHSc, University of Turku
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: NTSF2016
Record Dates: First submitted 2016-03-14; First posted 2016-03-24 (Estimated); Last update posted 2016-10-26 (Estimated); Status verified 2016-10

CONDITIONS: Smoking Prevention
Keywords: Games; Adolescent; Health education; Smoking; Health literacy
MeSH Terms: conditions — Health Education; Smoking

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (3):
- Health game group (Experimental): Participants in this arm will receive the health game intervention including both 20 minutes guided training session at school and 2 weeks free usage of the health game during free time.
  Interventions: Behavioral: Health game
- Web page group (Sham Comparator): Participants in this arm will receive the web page intervention including both 20 minutes guided training session at school and 2 weeks free usage of the web page during free time.
  Interventions: Behavioral: Web page
- Group with no intervention (No Intervention): The participants in this arm will receive no intervention.

INTERVENTIONS:
Behavioral: Health game — Health game intervention consists of 20 minutes guided training session with the health game at school and 2 weeks free usage of the health game via own smart phone or tablet computer during free time. The health game includes textual information about the consequences of tobacco use, but also visualized elements that aim at supporting understanding of the information, and motivation and ability to use the information in daily life situations. The visualized content is presented in a format of a game including tasks, rules, goals, rewards and opponents. There are also sound effects and background music included in the game.
  Arms: Health game group
Behavioral: Web page — Web page intervention consists of 20 minutes guided training session with the web page at school and 2 weeks free usage of the web page via own smart phone or tablet computer during free time. The web page includes textual information about the consequences of tobacco use, but also visualized elements that aim at supporting understanding of the information, and motivation and ability to use the information in daily life situations. The visualized elements are presented with pictures and video clips. These visualized elements do NOT contain game elements (NO activating tasks, rules, goals, rewards or opponents). The video clips contain sound effects, but no background music.
  Arms: Web page group

SUMMARY:
This feasibility study evaluates acceptability and preliminary effectiveness of a digital health game as an intervention supporting tobacco-related health literacy in 10- to 13-year-old early adolescents. One third of the study participants will receive the health game, on third a web page with similar content and one third will act as a control group without intervention.

ELIGIBILITY:
Inclusion Criteria:

* Goes to school at 4th, 5th or 6th grade
* Understands and can communicate either in Finnish, Swedish or English
* Has daily access to either a smart phone or tablet computer during free time

Exclusion Criteria:

* Takes part to specialized education

Ages: 10 Years to 13 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 151 (Actual)
Dates: Start 2016-03; Primary Completion 2016-06 (Actual); Study Completion 2016-06 (Actual)

PRIMARY OUTCOMES:
Change in anti-smoking self-efficacy | At baseline and at 2 weeks
  Assessed with Anti-smoking self-efficacy scale (ASSES)

SECONDARY OUTCOMES:
Change in smoking outcome expectations | At baseline and at 2 weeks
  Assessed with Smoking Outcome Expectation scale (SOES)
Change in attitudes towards tobacco use questionnaire scores | At baseline and at 2 weeks
  Assessed with a 4 point likert-scale questionnaire
Change in tobacco use-related motives questionnaire scores | At baseline and at 2 weeks
  Assessed with a 4 point likert-scale questionnaire
Actual use of the intervention | During 2 weeks period
  Actual use of the intervention is tracked with log files
Self-assessed interest towards the intervention | At 2 weeks
  Assessed with a 4 point likert-scale questionnaire

CONTACTS AND LOCATIONS:
Locations (1):
- Primary schools (n=6), Three Cities, Southwest Finland, Finland